CLINICAL TRIAL: NCT06871345
Title: Evaluation of the Links Between Perimenstrual Symptoms and Emotional Dysregulation in Autistic People: Ecological, Subjective, Cognitive and Physiological Approach.
Brief Title: Perimenstrual Symptoms and Emotional Dysregulation in Autism
Acronym: MEDEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9499; 2024-A02269-38 (Other: ANSM)
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Borderline Personality Disorder BPD
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Mental Status and Dementia Tests; Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy voluntary group (Active Comparator): 20 menstruating women with a regular menstrual cycle that lasts between 25 and 35 days, not using hormonal contraception and without a psychiatric and/or neurological diagnosis.
  Interventions: Other: Semi-structured interviews SCID; Other: Self-report questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA)
- Autism female patients group (Experimental): 20 female patients with a diagnosis of Autism Spectrum Disorder (ASD), according to DSM-5 criteria.
  Interventions: Other: Semi-structured interviews SCID; Other: Self-report questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA)
- Group of female patients with BPD (Experimental): 20 female patients with a diagnosis of BPD, according to DSM-5 criteria.
  Interventions: Other: Semi-structured interviews SCID; Other: Self-report questionnaires; Other: Cognitive assessment; Other: Momentary Ecological Assessment (EMA)

INTERVENTIONS:
Other: Semi-structured interviews SCID — Structured Clinical Interview for DSM-5 Personality Disorder (SCID) :
  The SCID is a 90-item semi-structured interview, covering all 10 categories of personality disorder as described in the DSM-5. Each item is rated on a three-point scale: "absent", "subclinical level" and "present".
Other: Self-report questionnaires — Participants will complete a battery of self-report questionnaires, assessing emotional dysregulation (including SRD, the primary endpoint), childhood adversity, anxiety, depression, and premenstrual symptoms.
Other: Cognitive assessment — Cognitive assessment, coupled with the recording of physiological parameters (Biopac).
  Participants will complete a battery of neuropsychological tests targeting emotional processes. These tests will make it possible to evaluate the hot component of executive functioning, i.e. specifically involved in the processing of socio-emotional information. Autobiographical verbal fluences and the emotional Hayling test will be used to measure initiation and inhibition processes, respectively.
Other: Momentary Ecological Assessment (EMA) — A momentary ecological evaluation protocol will be proposed between visits V1 and V4 in order to assess the emotional and symptomatic dynamics in a context of daily life. During two menstrual cycles, subjects will be invited, via their smartphone, to take daily semi-random readings (indicated by SMS) of their subjective (4 times/day), but also spontaneous emotional experiences

SUMMARY:
Emotional dysregulation (ED) is defined as difficulties in modulating the experience and expression of emotions, which are characterized by a particularly marked reactivity, intensity and duration.

In order to improve the understanding of ED, its consequences in autistic women, and to be able to offer them appropriate treatments, it seems crucial to investigate the links between ED, adversities experienced during childhood and premenstrual dysphoric symptoms.

This study aims to characterize the variability of ED along a menstrual cycle by measuring it in a real-life ecological context. The variability of ED will be compared to that of women with borderline personality disorder BPD and that of women without psychiatric disorders.

ELIGIBILITY:
Inclusion criteria:

Common Inclusion Criteria for Healthy Patients and Volunteers:

* Female aged 18 to 45;
* Woman with regular menstrual cycles (variations in duration, measured between the shortest menstrual cycle) and the longest cycle, remain strictly less than 7 days) between 25 and 35 days;
* Woman without hormonal contraception (or NON-hormonal copper IUD) or who has stopped contraception for more than 3 months (and does not wish to take it again);
* Woman with a smartphone with an internet connection;
* Woman able to understand the objectives and risks of the research and to give informed, dated and signed consent;
* Woman affiliated to a social protection health insurance scheme, beneficiary or beneficiary.

Patient-specific inclusion criteria:

* Patient with a diagnosis of Autism Spectrum Disorder without intellectual disability (ASD), according to the criteria of the DSM-5 OR
* Patient with a diagnosis of BPD, according to DSM-5 criteria

Exclusion criteria:

Non-inclusion criteria common to healthy patients and volunteers:

* Taking hormonal treatment or synthetic steroids;
* Woman using hormonal contraceptives (pill, patch, hormonal IUD, vaginal ring, implant, intramuscular injection);
* Pregnancy or breastfeeding on the declaration of the person for less than 3 months;
* Desire to become pregnant within 3 months of inclusion;
* Endocrinopathies (in particular clinical signs of hyperandrogenism) or untreated gynaecological pathologies that may influence menstrual cycles and/or ovulation;
* Participation in another study that may interfere with the study;
* Inability to give the person informed information (person in an emergency or life-threatening situation);
* Woman under judicial protection;
* Woman under guardianship or curatorship;
* Woman hospitalized for a period > 24 hours

Patient-specific non-inclusion criteria:

* Patient with a diagnosis of psychotic disorder;
* Patient with a diagnosis of severe substance use disorder, i.e., presence of 6 or more symptoms;
* Patient with a diagnosis of bipolar disorder type I or II or cyclothymia;
* Patient with a diagnosis of co-occurring ASD and BPD;
* Patient with an intellectual disability (IQ ≤ 70);
* Patient with neurological comorbidity (e.g., acquired brain injury);
* Patient on treatment that alters physiological response (heart rhythm, e.g., beta-blockers).

Non-inclusion criteria specific to healthy volunteers:

* Woman with a psychiatric, neurodevelopmental or neurological history;
* Woman on psychotropic therapy or treatment that modifies physiological parameters (e.g., beta-blockers).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients and female volunteers
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
The links between emotional dysregulation and premenstrual dysphoric symptoms in autistic women compared to women with borderline personality disorder and women without a diagnosed psychiatric disorder (healthy volunteers). | 3 months
  Comparison between groups (autistic people, people with BPD, people without disorders) of the intensity of ED assessed using self-report questionnaires according to the phase of the menstrual cycle (follicular phase, luteal phase and late luteal phase).

SECONDARY OUTCOMES:
The impact of the menstrual cycle on emotional manifestations | 3 months
  Correlation and mediation between scores on the emotional dysregulation (Emotional Regulation Scale 16, Shortened Scale of Emotional Dysregulation, Alexithymia Scale, Flexible Regulation of Emotional Expression Scale), childhood adversity and premenstrual dysphoric symptoms scales and Daily recording of the intensity of difficulties.
The impact of the menstrual cycle on cognitive manifestations | 3 months
  Correlation and mediation between scores on the emotional dysregulation (Emotional Regulation Scale 16, Shortened Scale of Emotional Dysregulation, Alexithymia Scale, Flexible Regulation of Emotional Expression Scale), childhood adversity and premenstrual dysphoric symptoms scales and Daily recording of the intensity of difficulties.
The impact of the menstrual cycle on behavioral manifestations | 3 months
  Correlation and mediation between scores on the emotional dysregulation (Emotional Regulation Scale 16, Shortened Scale of Emotional Dysregulation, Alexithymia Scale, Flexible Regulation of Emotional Expression Scale), childhood adversity and premenstrual dysphoric symptoms scales and Daily recording of the intensity of difficulties.
Subjective differences in real-life emotional experience between ASD, BPD, and healthy volunteers | 3 months
  Premenstrual dysphoric symptoms scores
Cognitive correlates of emotional dysregulation by phase of the menstrual cycle | 3 months
  Comparison of Suicidal Ideation Scale scores in the follicular, luteal, and mid-luteal phases of the menstrual cycle
The concordance between subjective, physiological and cognitive measures of emotional dysregulation, assessed in daily life, in ASD, BPD and healthy volunteers | 3 months
  Comparison of scores on the scales assessing emotional dysregulation, List of Borderline Symptoms 23, autistic traits (AQ), Depression, Anxiety and Stress Scale (EDAS-21) and depressive traits (EDAS-21, BDI) in the follicular phase and the late luteal phase of the menstrual cycle.
The concordance between cognitive and physiological measures of emotional dysregulation, assessed in consultation, in autistic people compared to people with BPD and healthy volunteers | 3 months
  Comparison of the frequency of emotional responses observed in a real-life context (ecological momentary assessment - EMA, according to the phase of the menstrual cycle (follicular phase, luteal phase and late luteal phase)
The association between subjective and cognitive measures of emotional dysregulation, assessed in consultation, in ASD compared to BPD and healthy volunteers | 3 months
  Comparison of the skin conductance recorded by the Empatica connected watch according to the phase of the cycle (follicular phase, luteal phase and late luteal phase)
Evaluate the intensity of dysphoric symptoms during two menstrual cycles | 3 months
  Comparison of performance at the proposed emotional Stroop task in daily life according to the phase of the menstrual cycle (follicular phase, luteal phase and late luteal phase
Understand the impact of these dysphoric symptoms during two menstrual cycles | 3 months
  Comparison of performance at the proposed emotional Stroop task in daily life according to the phase of the menstrual cycle (follicular phase, luteal phase and late luteal phase
The evolution of self-reported emotional dysregulation assessed in daily life during two menstrual cycles | 3 months
  Comparison in the follicular phase and in the late luteal phase of performances in the emotional Hayling.
The evolution of the emotional experience, assessed in daily life, during two menstrual cycles | 3 months
  Comparison of the evolution of the emotional experience between the three groups (autistic women, women with borderline personality disorder and control group
The evolution of physiological emotional responses, assessed in daily life and in consultation, during two menstrual cycles | 3 months
  Comparison of the evolution of physiological emtional reponses between the three groups (autistic women, women with borderline personality disorder and control group)
The evolution of cognitive functioning underlying emotional dysregulation, over the course of two menstrual cycles | 3 months
  Comparison of the evolution of cognitive functioning underlying emotional dysregulation between the three groups (autistic women, women with borderline personality disorder and control group)
The concordance between cognitive and physiological measures of emotional dysregulation, assessed in consultation, in autistic people compared to people with BPD and healthy volunteers | 3 months
  Comparison of the intensity of emotional responses observed in a real-life context (ecological momentary assessment - EMA, according to the phase of the menstrual cycle (follicular phase, luteal phase and late luteal phase)
The concordance between cognitive and physiological measures of emotional dysregulation, assessed in consultation, in autistic people compared to people with BPD and healthy volunteers | 3 months
  Comparison of the variability of emotional responses observed in a real-life context (ecological momentary assessment - EMA, according to the phase of the menstrual cycle (follicular phase, luteal phase and late luteal phase)
The association between subjective and cognitive measures of emotional dysregulation, assessed in consultation, in ASD compared to BPD and healthy volunteers | 3 months
  Comparison of the body temperature recorded by the Empatica connected watch according to the phase of the cycle (follicular phase, luteal phase and late luteal phase)
The association between subjective and cognitive measures of emotional dysregulation, assessed in consultation, in ASD compared to BPD and healthy volunteers | 3 months
  Comparison of the heart rate) recorded by the Empatica connected watch according to the phase of the cycle (follicular phase, luteal phase and late luteal phase)
The evolution of self-reported emotional dysregulation assessed in daily life during two menstrual cycles | 3 months
  Comparison in the follicular phase and in the late luteal phase of performances in a negative priming task.
The evolution of self-reported emotional dysregulation assessed in daily life during two menstrual cycles | 3 months
  Comparison in the follicular phase and in the late luteal phase of performances in a heart rhythm detection task proposed for consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa WEINER, Professor, Principal Investigator — Department of Psychiatry II Psychiatry, Mental Health and Addiction Medicine, University Hospitals of Strasbourg